CLINICAL TRIAL: NCT06414538
Title: The Effect Of Digital Mind Map Technique On Learning In Midwifery Students
Brief Title: The Effect of Digital Mind Map and Midwifery Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayla Ergin (Other)
Responsible Party: Sponsor-Investigator, Ayla Ergin, Professor Dr., Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ayla-2
Record Dates: First submitted 2024-03-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Education
Keywords: Digital mind; learning tool; midwifery; student success; motivation; family planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Mind Map Technique (Experimental): Students determined as a result of randomization will be given a pre-test before entering the "Family Planning"course planned according to the academic calendar. The planned topics will be explained using the prepared digital mind maps technique.
  Interventions: Other: Digital Mind Map Technique
- Classic Method Group (Active Comparator): The determined topics will be explained to the students in the control group using the classical method. Students' knowledge level will be measured with knowledge tests.
  Interventions: Other: Classic Method Group

INTERVENTIONS:
Other: Digital Mind Map Technique — Students determined as a result of randomization will be given a pre-test before entering the "Family Planning" course planned according to the academic calendar. The determined topics will be explained to the students using the digital mind map technique. A post-test will be administered to the students 1 week after the end of the subject and a satisfaction survey of the digital mind map technique will be administered. Permanence test will be applied 35 days after the last test application.
  Arms: Digital Mind Map Technique
Other: Classic Method Group — After the students in the control group are determined, a pre-test will be conducted before the subject is given training. The same knowledge test will be repeated as a final test after students have received classical course training and completed the subject. Students will be given a retention exam 35 days after the last exam. After the retention test application, the mind map method will be explained to the students in the control group and the determined topics of the course will be explained with the prepared digital mind map technique. In this way, all students participating in the study will also have access to the additional educational materials used.
  Arms: Classic Method Group

SUMMARY:
This study was conducted to determine the effect of the digital mind map technique on the learning of midwifery students. The research will be carried out with Kocaeli University Midwifery 2nd year students. A meeting was held with students regarding extracurricular studies between 12 February and 16 February 2024, which is the beginning of the 2023-2024 academic year academic calendar of Kocaeli University. The research will be completed with 86 students in the mind map method group (n = 43) and the classical method (n = 43) group. Data will be collected through the participant information form, knowledge assessment survey on family planning, and satisfaction assessment survey of the narrative regarding the digital mind map. Three topics determined regarding family planning methods (oral contraceptives, condoms and intrauterine devices) were prepared by the researcher using the digital mind map technique. The participant information form and the knowledge evaluation survey on family planning were administered as a pre-test to the students who accepted the research at the first meeting. The mind map technique was first explained to the mind map method group. The topics were explained to the students in the mind map method group by the researcher and his advisor using the mind map technique and with materials prepared with the digital mind map technique. The classical method was explained to the classical method group by the researcher and his advisor. A posttest will be administered to both groups 1 week after the lecture. Again, 35 days after the lecture, the study will be completed by applying a permanence test to both groups and a student satisfaction survey to the experimental group. After the study, the mind map technique will be explained to all students in the classical method group who have completed the study, and the topics prepared with the digital mind map technique will be explained to the classical method group and reinforced. Statistical analysis of the data obtained as a result of the research will be carried out using the IBM Statistic 22.0 (IBM Corp., Armonk, NY, USA) program. Study data will be collected using appropriate statistical methods and the significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Primary aim: The research is to determine the effect of digital mind mapping technique on learning in midwifery students.

Hypotheses:

H0: There is no difference between the knowledge evaluation survey average scores of students in the mind map method group and the classical method group.

H1: There is a statistically significant difference between the knowledge evaluation survey score averages of students in the mind map method group and the classical method group.

H2: There is no statistically significant difference between the satisfaction and motivation of students in the mind map method group and the classical method group.

H3: There is a statistically significant difference between the satisfaction and motivation of students in the mind map method group and the classical method group.

This study was designed as a randomized controlled experimental study. The study will be carried out at Kocaeli University Faculty of Health Sciences between February 2024 and May 2024.

In order to facilitate data collection, the population of the research will consist of 86 second-year midwifery students of Kocaeli University Faculty of Health Sciences in the 2023-2024 academic year. The sample size was based on Ahmed et al.'s 2023 study in which the method of the digital mind map strategy was examined. The sample number of the study was calculated using the G*Power 3.1.9.2 program, and the mean, standard deviation and sample number values of the knowledge test scores of the groups in the relevant article (Ahmed M.M,, Ismail E.H., Abousoliman, A, 2023) were taken into account in the effect size calculation. In the experimental group, the mean and standard deviation values of the knowledge score are 13.32±3.69 and the number of samples is 113. In the control group, the mean and standard deviation values of the knowledge score are 11.51±2.76 and the number of samples is 128. By using the mean, standard deviation and sample number values of the relevant article, the effect size was calculated as 0.560. According to the result of 95% confidence (1-α), 80% test power (1-β), d = 0.560 effect size, the minimum number of samples to be taken in each group is 16 people, a total of 32 people should be examined. In order to increase the power of analysis, n = 16 (mind map method group: 16 and classical method group: 16) will be taken for each group in the study. The students included in the research will be divided into two groups by determining which group they will belong to from the website called "Random Team Generator", which is a random number generation program. Thus, each student's number and group number will be determined and recorded.

Randomization: The mother group will be determined from the random number generator site called "Random Lists". Students will be divided into two groups: mind map method and classical method group. Thus, the number of each student will be determined and recorded.

Research data will be collected using the Participant Information Form, the Knowledge Evaluation Survey on Family Planning and the Satisfaction Evaluation Survey of the Explanation on Digital Mind Map.

Participant Information Form: Participant information form was created as a result of literature review. This form includes questions such as the students' age, employment status, educational status of their parents, place of residence during their student years, and reasons for choosing the midwifery department.

Knowledge Evaluation Survey on Family Planning: It was prepared to measure students' learning levels with a survey consisting of 30 questions as a result of literature review. The minimum value that can be obtained from the survey will be calculated as 0 and the maximum value will be calculated as 30. It will be understood that the higher the score the students receive, the better their knowledge level.

Expression Satisfaction Evaluation Survey on Digital Mind Map: As a result of the literature review, a survey consisting of 25 questions was prepared to measure students' satisfaction levels with the mind map technique. There is no minimum and maximum value range. The survey has been prepared in a way that can be marked more than once and is open to interpretation..

Before the research, a pilot study will be conducted with second-year students of Sakarya University, Faculty of Health Sciences, Department of Midwifery. This pilot study will be carried out by the researcher using face-to-face interview technique between 12.02.2024-16.02.2024. Students will be asked not to share the study with other students or on social media platforms by signing a consent form and confidentiality agreement.

Participants will be informed that they can leave the study at any time and the study will be completed with voluntary participants. All students participating in the research will sign a confidentiality agreement and will be ensured not to share their work with other students or on platforms such as social media. A participant information form consisting of 15 questions will be applied to each student participating in the research, and a knowledge assessment survey on family planning consisting of 30 questions will be applied to the students as a pre-test to measure their knowledge after the training.

Randomization will be made among the students who agree to participate in the research, and two groups will be created: the mind map method and the classical method group. The presentation of the topics is planned between March and May 2024. The topics will be explained to the students in the mind map method group by the researcher together with his advisor, using the mind map technique. In the classical method group, the topics will be explained by the researcher together with his advisor using the classical method. One week after the lecture, a posttest knowledge assessment survey on family planning will be administered to both groups to measure the change in the students' knowledge levels. 35 days after this post-test exam, a knowledge evaluation survey on family planning will be administered to all students to measure the permanence of the subjects. In addition, a student satisfaction survey will be applied to the mind map method group to measure the satisfaction levels of the students. After the retention test is applied, the mind map technique will be explained to the students in the classical method group, and the topics prepared with the digital mind map technique will be explained to the classical method group and reinforced

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Between the ages of 18-30,
* Kocaeli University Faculty of Health Sciences Midwifery 2nd year student
* Students who are not absent

Exclusion Criteria:

* Those who want to leave the study for any reason,
* Leaving questionnaires incomplete,
* Students who have previously received training on family planning

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level | 4 weeks
  It will be applied as a pre-test with the Knowledge Evaluation Survey on Family Planning in order to determine the students' knowledge levels. It was prepared to measure students' learning levels with a survey consisting of 30 questions. The minimum value that can be obtained from the survey will be calculated as 0 and the maximum value will be calculated as 30. It will be understood that the higher the score the students receive, the better their knowledge level.
Knowledge Level | 8 weeks
  After the topics are explained, the final test of the Family Planning Knowledge Evaluation Survey will be applied to determine the students' knowledge levels. It was prepared to measure students' learning levels with a survey consisting of 30 questions. The minimum value that can be obtained from the survey will be calculated as 0 and the maximum value will be calculated as 30. It will be understood that the higher the score the students receive, the better their knowledge level.
Satisfaction levels of materials prepared with the digital mind map technique | 2 weeks
  In order to evaluate the materials prepared with the digital mind map technique of the students in the experimental group, a Satisfaction Evaluation Survey of the Expression on Digital Mind Map will be conducted. It is a survey consisting of 25 questions. There is no minimum and maximum value range. The prepared survey was prepared in a way that you could mark more than once and was open to interpretation.
Knowledge Level | 12 weeks
  It will be applied as a retention test of the Family Planning Knowledge Evaluation Survey to determine the students' knowledge levels. It was prepared to measure students' learning levels with a survey consisting of 30 questions. The minimum value that can be obtained from the survey will be calculated as 0 and the maximum value will be calculated as 30. It will be understood that the higher the score the students receive, the better their knowledge level.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Ergin, Prof. Dr., Principal Investigator — ergina@kocaeli.edu.tr; Sema Güneş Yanık, Graduate st, Study Chair — ebesemagunes@gmail.com
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)